CLINICAL TRIAL: NCT07178496
Title: Effect of Integrating Sleep Hygiene Techniques With Physiotherapy Exercise in Improving Sleep Quality and Disability in Patients With Chronic Neck Pain
Brief Title: Sleep Hygiene Plus Physiotherapy for Sleep and Disability in Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mosab ALdabbas, Assistant Professor, Al Zhar University, Gaza, Palestine _ Field physiotherapy Officer, International committee of the red cross, Gaza, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL Azhar university, GAZA STRI
Record Dates: First submitted 2025-08-27; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Neck Pain Musculoskeletal; Sleep Disturbances; Fatigue, Mental
Keywords: sleep quaity; sleep hygiene; neck pain
MeSH Terms: conditions — Neck Pain; Parasomnias; Mental Fatigue; Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group receive conventional Physiotherapy program (Experimental): Conventional Physiotherapy Program
  1. Treatment Frequency and Duration
     Frequency: 3 sessions per week
     Duration: 8 weeks
     Session length: 45-60 minutes
  2. Hot Pack Application (10-15 minutes)
  Purpose: Reduce pain, improve soft-tissue extensibility, and prepare muscles for exercise.
  Procedure:
  Moist hot pack applied to the cervical region.
  Temperature: 40-45°C (comfortable warmth, checked to avoid burns).
  Duration: 10-15 minutes with adequate towel layers.
  Neck Endurance and Strength Training (30-40 minutes)
  Interventions: Other: conventional physiotherapy program
- Group receive conventional Physiotherapy program plus sleep hygiene technique (Experimental): Exercise
  and
  1. Delivery Method
     Initial Education Session:
     A 45-minute one-on-one session with a physiotherapist or trained researcher.
     Delivered face-to-face using visual aids (slides, posters, printed guide).
     Explains what sleep hygiene is, why it matters in chronic neck pain, and how to apply each strategy.
     Follow-up Sessions:
     Weekly 15-20-minute reinforcement sessions (in-person or by phone/video call).
     Used to review progress, clarify doubts, troubleshoot barriers, and adjust advice if necessary.
     Written Materials:
     A patient booklet summarizing all recommendations in simple language, including diagrams of neck-friendly sleeping postures.
     A daily sleep diary to track bedtime, wake time, naps, and perceived sleep quality.
  2. Program Content A. Regular Sleep-Wake Timing
  Go to bed at the same time every night and wake at the same time every morning, even on weekends.
  Use alarms only for waking, not for forcing sleep onset.
  Limit naps to <30 minutes, no later than 4
  Interventions: Other: Sleep Hygiene Techniques
- control (Other): advices and home program
  Interventions: Other: Control arm

INTERVENTIONS:
Other: Sleep Hygiene Techniques — Sleep Hygiene Techniques
  The sleep hygiene program includes education and behavioral strategies to promote healthier sleep patterns, delivered alongside physiotherapy exercises. Key components are:
  Regular Sleep-Wake Schedule
  Encourage patients to maintain consistent bedtime and wake-up times, even on weekends.
  Avoid excessive time in bed when not sleeping.
  Optimizing the Sleep Environment
  Ensure a quiet, dark, and cool bedroom (18-22°C).
  Use supportive pillows to maintain neutral cervical alignment and reduce neck strain.
  Remove distractions such as TVs, mobile phones, and bright lights.
  Pre-Sleep Routine
  Establish a relaxing wind-down routine (e.g., gentle stretching, breathing exercises, reading).
  Avoid mentally stimulating activities or heavy problem-solving before bedtime.
  Limiting Stimulants and Alcohol
  Avoid caffeine, nicotine, and alcohol at least 4-6 hours before bedtime.
  Avoid heavy meals close to bedtime; a light snack is acceptable if hungry.
  Daytime Habits t
  Arms: Group receive conventional Physiotherapy program plus sleep hygiene technique
Other: conventional physiotherapy program — Conventional Physiotherapy Program
  1. Treatment Frequency and Duration
     Frequency: 3 sessions per week
     Duration: 8 weeks
     Session length: 45-60 minutes
  2. Hot Pack Application (10-15 minutes)
     Purpose: Reduce pain, improve soft-tissue extensibility, and prepare muscles for exercise.
     Procedure:
     Moist hot pack applied to the cervical region.
     Temperature: 40-45°C (comfortable warmth, checked to avoid burns).
     Duration: 10-15 minutes with adequate towel layers.
  3. Neck Endurance and Strength Training (30-40 minutes)
  Arms: Group receive conventional Physiotherapy program
Other: Control arm — only advices and home advices
  Physiotherapy Advice for Patients with Neck Pain
  Adhere to Your Exercise Program
  Perform the prescribed neck strengthening and endurance exercises daily.
  Focus on quality over quantity-slow, controlled movements are more effective.
  Maintain Correct Posture During All Activities
  Keep your neck in a neutral position whether sitting, standing, or walking.
  Incorporate Frequent Micro-Breaks
  Every 30-45 minutes, pause to gently move and stretch your neck and shoulders.
  Small posture corrections throughout the day prevent stiffness.
  Use Heat Before Exercise if Stiff or Painful
  Apply a hot pack for 10-15 minutes before exercises to relax muscles.
  Avoid prolonged or excessive heat application.
  Stay Active - Avoid Prolonged Rest
  Light physical activity (walking, cycling, gentle mobility work) helps recovery.
  Bed rest should be avoided unless pain is severe.
  Practice Relaxation and Breathing C
  Arms: control

SUMMARY:
This study investigates the effectiveness of a combined intervention that integrates sleep hygiene education with physiotherapy exercises in patients suffering from chronic neck pain. Chronic neck pain is often associated with both musculoskeletal dysfunction and secondary sleep disturbances, which in turn may exacerbate pain perception, fatigue, and disability. Traditional physiotherapy exercise programs focus primarily on improving cervical mobility, muscle strength, and postural control, but they do not typically address sleep-related problems that can hinder recovery.

The intervention in this study consists of two main components:

Physiotherapy Exercise Program - A structured regimen targeting cervical spine mobility, deep cervical flexor strengthening, scapular stabilization, and postural correction. These exercises aim to reduce pain, restore function, and improve overall physical performance.

Sleep Hygiene Education - A structured educational module covering principles of healthy sleep habits, including maintaining consistent sleep-wake schedules, creating an optimal sleep environment, limiting stimulants before bedtime, and adopting relaxation strategies to promote better sleep initiation and maintenance.

By combining these approaches, the intervention addresses not only the physical impairments associated with chronic neck pain but also the psychosocial and behavioral factors contributing to poor sleep quality.

Outcome Measures:

Primary Outcomes: Sleep quality, assessed using validated tools such as the Pittsburgh Sleep Quality Index (PSQI).

Secondary Outcomes: Disability and functional limitations, measured by the Neck Disability Index (NDI), along with pain intensity assessed using a Visual Analog Scale (VAS).

Fatigue will be assessed by fatigue inventory index

Study Hypothesis: The combined intervention of sleep hygiene education and physiotherapy exercise will lead to greater improvements in sleep quality and reductions in disability and fatigue compared to physiotherapy exercise alone.

Clinical Significance: If effective, this integrative approach may provide a cost-effective, non-pharmacological management strategy for patients with chronic neck pain, targeting both physical and behavioral contributors to their condition.

ELIGIBILITY:
Inclusion Criteria

Participants will be eligible for the study if they meet the following conditions:

1. Adults aged 20-55 years.
2. Clinical diagnosis of chronic neck pain, defined as symptoms persisting for more than 3 months.
3. Poor sleep quality, indicated by a Pittsburgh Sleep Quality Index (PSQI) score >5.
4. Willingness to participate and comply with both the physiotherapy and sleep hygiene intervention program.
5. Ability to provide informed consent.

Exclusion Criteria

Participants will be excluded if any of the following conditions are present:

1. History of cervical spine trauma, surgery, or fracture within the past 6 months.
2. Severe depression or anxiety, defined by scores above the severe threshold on the Hospital Anxiety and Depression Scale (HADS).
3. Neurological disorders affecting neck function (e.g., cervical radiculopathy, myelopathy).
4. Other musculoskeletal disorders causing significant neck or shoulder pain.
5. Sleep disorders unrelated to neck pain (e.g., obstructive sleep apnea, restless legs syndrome, narcolepsy), whether diagnosed or suspected.
6. Ongoing pharmacological treatments that may significantly affect sleep (e.g., sedatives, hypnotics), unless the patient has been on a stable dose for >3 months.

6 Uncontrolled systemic illnesses such as diabetes, cardiovascular disease, or cancer.

7 Pregnancy.

8 Participation in any recent physiotherapy program targeting neck pain within the last 3 months.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
sleep quality | pre and 8 weeks post interventions as well as 8 weeks follow up
  Pittsburgh Sleep Quality Index (PSQI):
  The PSQI is a widely used and validated self-reported questionnaire designed to assess sleep quality and disturbances over a 1-month period. It consists of 19 individual items that generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored on a 0-3 scale, and the sum of these components yields a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality. A global score greater than 5 is typically used to distinguish poor sleepers from good sleepers. The PSQI provides a comprehensive overview of both qualitative and quantitative aspects of sleep, making it a suitable primary outcome measure in this study.
Disability | Pre, 8 weeks post PT intervention's and 8 weeks follow up
  Neck Disability Index (NDI):
  The NDI is a standardized, condition-specific outcome measure used to determine the level of disability in individuals with neck pain. It contains 10 items addressing pain intensity and the impact of neck pain on daily activities such as personal care, lifting, reading, concentration, work, driving, sleeping, and recreation. Each item is scored on a 0-5 scale, with the total score ranging from 0 to 50, which can then be expressed as a percentage. Higher scores reflect greater disability. The NDI is recognized as a reliable and valid tool for evaluating functional limitations and tracking treatment progress in patients with chronic neck pain.

SECONDARY OUTCOMES:
Pain | Pre, 8 weeks post PT and 8 weeks follow up
  Visual Analog Scale (VAS) for Pain:
  The VAS is a simple, validated tool used to measure pain intensity. It typically consists of a 10-centimeter horizontal line, with the left end representing "no pain" and the right end representing "worst imaginable pain." Patients are asked to mark a point along the line that best represents their perceived pain intensity at the time of assessment. The score is determined by measuring the distance in centimeters from the left end of the line to the patient's mark, yielding a score between 0 and 10. The VAS is highly sensitive to changes in pain over time and is widely used in clinical and research settings to evaluate treatment effectiveness.
Fatigue | Pre, 8 weeks post PT interventions, and 8 weeks follow up
  Fatigue Severity Scale (FSS):
  The Fatigue Severity Scale is a self-reported questionnaire designed to assess the severity and impact of fatigue on daily functioning. It consists of nine statements that evaluate how fatigue interferes with motivation, exercise, physical functioning, and social life. Each statement is rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). The mean of all item scores is calculated, with higher scores indicating greater fatigue severity. The FSS is a reliable and valid measure, particularly relevant in chronic pain populations, as fatigue is a common and often overlooked symptom that contributes significantly to reduced quality of life.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gupta CC, Sprajcer M, Johnston-Devin C, Ferguson SA. Sleep hygiene strategies for individuals with chronic pain: a scoping review. BMJ Open. 2023 Feb 2;13(2):e060401. doi: 10.1136/bmjopen-2021-060401. PMID 36731933